CLINICAL TRIAL: NCT04065165
Title: Randomized Phase III Clinical Trial of Lanreotide Combined With Telotristat Ethyl or Placebo for the First-line Treatment in Patients With Advanced Well Differentiated Small Intestinal Neuroendocrine Tumours (siNET) With Highly-functioning Carcinoid Syndrome
Brief Title: Lanreotide Combined With Telotristat Ethyl or Placebo for the First-line Treatment in Patients With Advanced Well Differentiated Small Intestinal Neuroendocrine Tumours (siNET) With Highly-functioning Carcinoid Syndrome
Acronym: TELEFIRST
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EORTC-1715-GITCG
Record Dates: First submitted 2019-08-14; First posted 2019-08-22 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Small Intestinal NET; Carcinoid Heart Disease
Keywords: intestinal NET; carcinoid syndrome; somatostatin analogues; tryptophan hydroxylase inhibitor
MeSH Terms: conditions — Carcinoid Heart Disease; Serotonin Syndrome | interventions — telotristat ethyl; lanreotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Lanreotide 120 mg q4w Telotristat Ethyl 250 mg TID
  Interventions: Drug: Telotristat Ethyl; Drug: Lanreotide
- Control arm (Placebo Comparator): Lanreotide 120 mg q4w Placebo TID
  Interventions: Drug: Lanreotide

INTERVENTIONS:
Drug: Telotristat Ethyl — 250 mg TID orally
  Other Names: Xermelo
  Arms: Experimental arm
Drug: Lanreotide — 120 mg Q4W deep subcutaneous injection in the superior external quadrant of the buttock or in the upper outer thigh
  Other Names: Somatuline

SUMMARY:
This is a randomized phase III clinical trial of Lanreotide combined with Telotristat ethyl or placebo for the first-line treatment in patients with advanced well differentiated small intestinal neuroendocrine tumours (siNET) with highly-functioning carcinoid syndrome to test whether telotristat ethyl plus lanreotide is more effective than placebo plus lanreotide in reducing the number of daily bowel movements.

In addition, the study allows evaluation of the biochemical response (5-HIAA and chromogranin-A), the reduction in the number of daily cutaneous flushing episodes, the improvement in abdominal pain/discomfort, health-related quality of life, improvement in gastro-intestinal and endocrine symptoms, changes in emotional functioning, the impact of discontinuation of telotristat ethyl/placebo on HRQOL and symptoms, and the safety and toxicity of the treatment.

Patients will enter into a screening/run-in period of 1 week to establish baseline characteristics and symptomatology. The baseline assessment of daily bowel movement, as assessed in an electronic diary, will be averaged over the run-in period.

Following the screening/run-in period, patients will be randomly assigned (1:1) to either the control arm or the experimental arm for 12 months. Randomization will be stratified according to the grade of tumour differentiation (grade 1 vs. grade 2) and by baseline number of bowel movements per day (4-6 versus >6). A total of 94 patients will be randomly assigned (1:1) to either arm.

Upon randomization, all patients will enter the 12-month treatment period with lanreotide + telotristat ethyl/placebo (blinded). In the experimental arm, patients will receive the deep subcutaneous injection of lanreotide (120 mg) every 28 days and 250 mg orally three times daily (TID) of telotristat ethyl for 12 months. In the control arm, patients will receive the deep subcutaneous injection of lanreotide every 28 days (120 mg) and placebo orally TID for 12 months.

After completion of a minimum of 6 months on randomized blinded-treatment, the protocol allows for patients on treatment with telotristat ethyl/placebo to be unblinded in the event of "lack of symptom control". Unblinding due to "lack of symptom control" can happen at any time between 6 and 12 months of the blinded-treatment period. After unblinding, patient will interrupt protocol treatment and will be further treated as per clinician discretion.

All patients will be unblinded after a maximum of 12 months on randomized blinded-treatment.

After a follow-up of 12 months, patients will go off study except patients with carcinoid heart disease. Patients off study will be further treated as per clinician discretion.

Patients with carcinoid heart disease will continue open-label treatment on study (lanreotide + telotristat ethyl or lanreotide alone according to what they were receiving at unblinding at 12 months) for 4 additional years (open-label extension period). Patients with carcinoid heart disease who discontinue protocol treatment before 12 months will also enter the extension period for additional follow-up. Additional follow-up will last 4 years for these patients and will include 6-monthly cardiological assessments.

All efficacy analyses will be conducted in the Intention-to-treat population as primary analyses i.e. all 94 randomized patients will be analyzed in the arm they were allocated by randomization. Safety analyses will be performed on the Safety population i.e. on all patients who have received at least one dose of the study drugs.

The translational research projects include blood metabolite discovery and targeted assays to find new biomarker candidates of response to Telotristat.

Human biological material that will be collected for translational research purpose:

* whole blood, plasma and serum at baseline, 4 hours after first dose, 4 weeks, 12 weeks and at end of treatment visit with telotristat/placebo (due to end of study, disease progression or lack of benefit)
* archival tissue samples (formalin-fixed paraffin-embedded) will be retrieved for all patients at study entry. In addition, one EDTA blood tube of whole blood (10 ml) at baseline, 12 weeks and end of treatment (EOT visit) might be also collected for not yet pre-defined and further translational research.

Quality of life will be assessed with the EORTC Quality of Life Questionnaire (QLQ-C30) version 3, together with the QLQ-GI.NET21 specific module designed for Neuroendocrine Tumours. The computer-adaptive testing (CAT) diarrhea scale will also be used. The baseline questionnaires must be completed during the screening period and before randomization. Subsequent questionnaires are completed at 4 weeks, 12 weeks, 24 weeks, 36 weeks and 52 weeks. Once a patient has stopped treatment, HRQoL data collection for that patient is required 1 month (28-35 days) after protocol treatment discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed well-differentiated (grade 1 or grade 2) neuroendocrine tumour from small bowel primary (or unknown primary suspected to be of small bowel origin) as per WHO / ENETS classification
* Advanced disease (locally advanced, metastatic or recurrent, according to TNM staging version 8 or ENETS latest classification), not amenable for curative surgery
* No previous systemic treatment for the advanced neuroendocrine tumour (including somatostatin analogue)
* Highly functioning carcinoid syndrome, defined as:

  * Mean ≥4 bowel movements per day; patients will have a one-week run-in screening period for recording of frequency and consistency of diarrhea (Only those who complete the one-week run-in screening period and are ≥6 days out of 7 compliant with diary entries will be considered eligible and randomized).

And

- Serum, plasma or urine 5-HIAA levels ≥2 ULN (within 28 days of study entry)

* Age ≥18 years (no upper limit) and life expectancy >3 months
* Adequate haematological, hepatic and renal laboratory values:
* Neutrophils >1500 cells/mm3
* Platelets >75,000 cells/mm3
* Hemoglobin (Hgb) >9 g/dL for males and >8 g/dL for females
* Aspartate transaminase (AST) and alanine aminotransferase (ALT): <2.5 x upper limit of normal (ULN) if patient does not have documented history of hepatic metastases or <5.5 x ULN if patient has documented history of hepatic metastases
* Total bilirubin ≤1.5 x ULN (unless patient has a documented history of Gilbert's Syndrome)
* Alkaline phosphatase (ALP) <5 x ULN, if total bilirubin is >ULN
* Serum creatinine <1.5 x ULN and with creatinine clearance > 30 ml/min as calculated with MDRD Formula
* Women of child bearing potential (WOCBP) MUST have a negative serum pregnancy test within 3 days prior to the first dose of study treatment.
* Unless child bearing potential has been terminated by surgery / radical radiotherapy, women of childbearing / reproductive potential should use highly effective birth control measures, during the study treatment period and for at least 30 days after the last study treatment and then according to the investigator recommendation or national/institutional guideline. A highly effective method of birth control is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly.
* Female subjects who are breast feeding should discontinue nursing prior to the first dose of study treatment and until 5 months months after the last study treatment.
* Before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Patients who are planned to be treated with other anti-tumour treatment (e.g. chemotherapy, liver embolization, Peptide Receptor Radionuclide Therapy (PRRT)) at the time of the study entry.
* Major surgery defined as procedures requiring general anesthesia or major regional anesthesia within 8 weeks prior to registration.
* Administration of any investigational therapeutic agent prior to registration (investigational imaging tracers are allowed).
* Patients who received any previous systemic treatment for carcinoid syndrome or tumour control (including SSA); previous use of anti-diarrheal medication such as loperamide or codeine is allowed.
* Patient with diarrhea and/or flushing due to any cause other than the neuroendocrine tumour such as fat malabsorption, bile acid malabsorption, enteric pathogens (parasites or clostridium difficile), short bowel syndrome (SBS) or malignancy.
* Allergy / history of hypersensitivity reaction to any of the treatment components.
* Any evidence of severe or uncontrolled systemic disease which, in the view of the investigator, makes it undesirable for the patient to participate in the trial.
* Patients with end-stage renal disease requiring dialysis.
* Patients with severe hepatic impairment (Child-Pugh score C).
* Patients with known rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.
* Any patient with a medical or psychiatric condition that impairs their ability to give informed consent.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Inclusion/Exclusion Criteria for long-term follow-up for carcinoid heart disease (assessed locally)

* Patients diagnosed with carcinoid heart disease during the baseline or 12-month treatment period will be eligible
* Patients with suspected carcinoid heart disease but with poor/limited transthoracic echocardiogram windows, will not be eligible for long-term carcinoid heart disease follow-up
* Patients with moderate/severe valvular heart disease secondary to any pathology other than carcinoid heart disease (as classified by the ESC valvular heart disease guidelines10) are not eligible
* Patients with any pre-existing right sided heart disease such as arrythmogenic ventricular cardiomyopathy and patients with pre-existing atrial or ventricular arrythmia are not eligible
* Patients with pre-existing cardiomyopathy (such as hypertrophic cardiomyopathy or dilated cardiomyopathy) are not eligible
* Patients with implanted cardiac devices (i.e. pacemakers or an implantable cardioverter defibrillator) are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Number of bowel movements (BMs) | 43 months after first patient in
  The change from baseline in the number of bowel movements (BMs) per day

SECONDARY OUTCOMES:
Urine/serum/plasma 5-HIAA and chromogranin-A | 43 months after first patient in
  Intrapatient change from baseline in urine/serum/plasma 5-HIAA and chromogranin-A
Number of daily cutaneous flushing episodes | 43 months after first patient in
  Change from baseline in the number of daily cutaneous flushing episodes.
Health Related Quality of Life (HRQoL) | 43 months after first patient in
  Quality of life will be assessed with the EORTC Quality of Life Questionnaire (QLQ-C30) version 3. Scale measures are: not at all; a little; quite a bit; very much.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Valle, Principal Investigator — The Christie NHS Foundation Trust, Manchester, UK; Angela Lamarca, Principal Investigator — The Christie NHS Foundation Trust, Manchester, UK